CLINICAL TRIAL: NCT01976611
Title: Safety and Efficacy of Botulinum Toxin Type A (BOTOX®) to Treat Chronic Migraine in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-139
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Migraine Disorders; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Patients who receive botulinum toxin Type A (BOTOX®) treatment for chronic migraine as per local standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A treatment for chronic migraine as per local standard of care in clinical practice.

SUMMARY:
This study is a Post-Marketing Surveillance study in Korea to evaluate the safety and efficacy of botulinum toxin Type A to treat Chronic Migraine in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with botulinum toxin Type A for chronic migraine in clinical practice.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with botulinum toxin Type A for chronic migraine in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Adverse Drug Reactions | 4 Years
Headache Impact Test-6 (HIT-6) Score Using a 5-Point Scale | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea